CLINICAL TRIAL: NCT01067404
Title: TIV Infant/Toddler Response Evaluation (TITRE)- Follow-up & Focus on Influenza B
Acronym: TITRE II
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: British Columbia Centre for Disease Control (Other Government)
Responsible Party: Dr. Danuta M. Skowronski, BC Centre for Disease Control
Other Study IDs: CIHR 200903CVC-203708/99971
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Influenza
Keywords: Influenza vaccines; Infant; Dose-Response relationship, immunologic
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 2008-09 study TIV recipients: Infants and toddlers who participated in earlier clinical trial (TITRE) to evaluate dosing (0.25mL versus 0.5mL) of trivalent influenza vaccine (TIV)
  Interventions: Biological: Trivalent inactivated influenza vaccine

INTERVENTIONS:
Biological: Trivalent inactivated influenza vaccine — 0.25mL dose of 2009-10 trivalent inactivated influenza vaccine (TIV)

SUMMARY:
Each winter, viruses belonging to two kinds of influenza A ("A/H1N1" & "A/H3N2") and two kinds of influenza B ("B/Yamagata" & "B/Victoria") can cause illness. The yearly influenza vaccine is designed to protect against both kinds of influenza A but only one or the other kind of influenza B. The vaccine is changed from year to year, meaning it may include one kind of B virus one year and the other kind another year. But because influenza is so hard to predict, sometimes the kind of B virus chosen for the vaccine may not match the kind that is causing illness. The National Advisory Committee on Immunization recommends that all infants and toddlers receive influenza vaccine to protect against their high rates of hospitalization. Infants/toddlers receiving influenza vaccine for the first time must get two doses (prime plus boost) to have a good antibody response. If they have ever before received a single dose of influenza vaccine, then they are recommended to receive only one dose each year afterwards. But we don't know how well previous doses of one kind of influenza B set the stage for good antibody response to a single dose of the other kind of influenza B. This study will try to answer that question in a group of infants/toddlers who last year received two doses of one kind of B virus ("Yamagata"), as part of another study. This year, we will give them a single dose of influenza vaccine that now contains the other kind of B virus ("Victoria") and see how much antibody they make to both kinds. About half these children received a higher amount of influenza vaccine in the previous year's study, so we will also compare their antibody levels on that basis. Since influenza B is an illness especially of children, understanding how to best protect infants/toddlers against both kinds of influenza B is important. This study will help us know if we need to design a new vaccine that not only includes both kinds of influenza A, but also both kinds of influenza B.

ELIGIBILITY:
Inclusion Criteria:

* Child previously participated in the TITRE I study;
* Child is healthy (stable chronic conditions acceptable) as established by health assessment interview and verbal history-directed health examination;
* Child has received the 2009 pandemic H1N1 influenza vaccine;
* Child is available and can complete all relevant procedures during the study period;
* Parent or legal guardian is available and can be reached by phone during the study period;
* Parent/guardian provides written informed consent;
* And, parent/guardian is fluent in English/French.

Exclusion Criteria:

* Child has already received the 2009-10 seasonal (TIV) influenza vaccine;
* Child has received immune globulin or other blood products within the prior six weeks;
* Child has received injected or oral steroids within prior six weeks;
* Child is or will be enrolled in any other clinical trial of a drug, vaccine or medical device during the study period;
* Or, child has a recently acquired health condition which, in the opinion of the investigator, would interfere with the evaluation or pose a health risk to the child.

Ages: 18 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants of earlier clinical trial (TITRE I); enrolled in winter 2008/09 as previously unimmunized infants and toddlers (6-23 months of age)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-02

PRIMARY OUTCOMES:
Immunogenicity based on CPMP criteria (seroprotection, defined as reciprocal HI titre equal to/greater than 40; seroconversion rate and factor) for B/Brisbane/60/2008(Victoria)-like and B/Florida/4/06(Yamagata)-like viruses | 4-6 weeks after receipt of TIV

CONTACTS AND LOCATIONS:
Overall Officials: Danuta M Skowronski, MD, Principal Investigator — BC Centre for Disease Control, Vancouver, Canada
Locations (3):
- Canada (3):
  - BC Centre for Disease Control, Vancouver, British Columbia
  - McGill University Health Centre - Vaccine Study Centre, Montreal, Quebec
  - Université Laval - Unité de recherche en santé publique, Québec, Quebec

REFERENCES:
- [Derived] Skowronski DM, Hottes TS, De Serres G, Ward BJ, Janjua NZ, Sabaiduc S, Chan T, Petric M. Influenza Beta/Victoria antigen induces strong recall of Beta/Yamagata but lower Beta/Victoria response in children primed with two doses of Beta/Yamagata. Pediatr Infect Dis J. 2011 Oct;30(10):833-9. doi: 10.1097/INF.0b013e31822db4dc. PMID 21857263